CLINICAL TRIAL: NCT05231668
Title: A Phase 1b, Single Ascending Dose, Randomized, Double-blind Study to Evaluate the Safety, Tolerability, and Activity of SAR439459 in Adults With Osteogenesis Imperfecta
Brief Title: Single Ascending Dose Study of SAR439459 in Adults With Osteogenesis Imperfecta (OI)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SAD17378; U1111-1269-6569 (Registry Identifier: ICTRP); 2024-511369-12-00 (Registry Identifier: CTIS); 2021-004914-21 (EudraCT Number)
Record Dates: First submitted 2022-01-31; First posted 2022-02-09 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR439459 (Experimental): Participants will receive a single dose of SAR439459
  Interventions: Drug: SAR439459
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR439459 — Powder for solution for infusion; IV infusion
  Arms: SAR439459
Drug: Placebo — Solution for infusion; IV infusion
  Arms: Placebo

SUMMARY:
SAR439459 is a human anti-Transforming growth factor β (TGFβ) monoclonal antibody. This phase 1 clinical study investigates the safety, tolerability, and activity of a single dose of SAR439459 in adult participants with OI.

Participants will receive a single IV dose of SAR439459 with safety, pharmacokinetic (PK), and pharmacodynamic (PD) assessments over 24 weeks.

There will be up to 3 dose cohorts. In addition to safety, tolerability, and PK assessments, bone mineral density (BMD) will be evaluated by dual-energy Xray absorptimetry (DXA) scan and a series of blood biomarkers will be monitored to document pharmacodynamic effects of the single dose of SAR439459.

DETAILED DESCRIPTION:
The duration of the study for all participants will be approximately 29 weeks:

* Up to 5 weeks from initiation of screening to dose administration
* Treatment on Day 1
* Follow-up and observation of safety and PD for 24 weeks
* Final study visit at Week 24

ELIGIBILITY:
Inclusion Criteria:

* Participants who are clinically categorized as Type I or IV osteogenesis imperfecta with a previously documented pathogenic genetic variant in human collagen type 1 alpha 1 gene (COL1A1) or human collagen type 1 alpha 2 gene (COL1A2).
* Participants who have experienced at least 1 bone fracture in the past 10 years OR 2 or more (≥2) fractures since the age of 18.
* Body weight ≥30.0 kg.
* Contraception for sexually active male participants or female patient; not pregnant or breastfeeding; no sperm donating for male participant.
* Signed written informed assent/consent.

Exclusion Criteria:

* Previously installed rods or metal hardware that would prevent bone mineral density evaluation of the lumbar spine (note: only two of the L1-L4 vertebrae are necessary for evaluation).
* History of moderate (25-40°) to severe (>40°) scoliosis assessed as Cobb angle (unless scoliosis does not impact assessment of bone mineral density in the lumbar vertebrae in the opinion of the investigator).
* Postmenopausal women who:

  * Are within 5 years of the onset of menopause (for example less than 5 years from their last menstruation or post-hysterectomy), however if the person has been on hormone replacement therapy for more than 1 year prior to enrollment, then they are eligible regardless of time from onset of menopause. The person must be willing to continue hormone replacement therapy throughout the study duration. OR
  * Were previously on hormone replacement therapy but have stopped within the past 5 years.
* History of treatment with denosumab, anti-sclerostin antibody, parathyroid hormone, bisphosphonates, or any other experimental therapy for OI within 6 months prior to any study baseline assessment.
* Known bleeding disorder.
* History of significant bleeding event that required hospitalization, surgery, or a blood transfusion that was possibly associated with increased bleeding tendency.
* Any major surgery within the last 28 days prior to investigational medicinal product (IMP) administration.
* Elective surgery or invasive procedure anticipated within 6 months after the IMP administration.
* Therapeutic doses of anticoagulants or antiplatelet agents (eg, 1 mg/kg bid of enoxaparin, 300 mg of aspirin daily, and 75 mg of clopidogrel daily or equivalent) within 7 days prior to the IMP administration.
* Any known central nervous system (CNS) or intraocular lesion that has a risk of bleeding.
* Prior history of skin cancers including melanoma, squamous cell carcinoma, or basal cell carcinoma.
* Clinically significant cardiac valvular disorder or symptomatic heart failure.
* Vitamin D (25-hydoxyvitamin D) <15 ng/dL; rescreening will be allowed after supplementation.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs)/treatment-emergent adverse events (TEAEs) | From baseline to Week 24

SECONDARY OUTCOMES:
Assessment of PK parameters: area under the curve (AUC) | From baseline to Week 24
Assessment of PK parameters: maximum serum concentration observed (Cmax) | From baseline to Week 24
Assessment of PK parameters: time to reach maximum concentration observed (tmax) | From baseline to Week 24
Titer of anti-SAR439459 antibodies (if detected) | From baseline to Week 24
Percent change from baseline in bone mineral density (BMD) | From baseline to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- United States (7):
  - UCLA Health_Site Number: 8400006, Los Angeles, California
  - Yale University - Site Number:8400007, New Haven, Connecticut
  - Indiana University School of Medicine_Site Number: 8400002, Indianapolis, Indiana
  - Kennedy Krieger Institute_Site number 8400004, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center Site Number : 8400010, Cincinnati, Ohio
  - Vanderbilt University Site Number : 8400011, Nashville, Tennessee
  - Baylor College of Medicine - Site Number:8400003, Houston, Texas
- Australia (2):
  - Westmead Hospital_Site Number :0360003, Westmead, New South Wales
  - Department of Medicine/ School of Clinical Sciences at Monash Health Monash University_246 Clayton Road_Site Number :0360002, Clayton, Victoria
- Canada (2):
  - Bone Research and Education Centre_Site Number :1240003, Oakville, Ontario
  - Toronto general Hospital_Site Number :1240002, Toronto
- France (2):
  - Hopital Edouard Herriot _Site Number :2500002, Lyon
  - Hopital Lariboisiere_Site Number :2500001, Paris

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: SAD17378 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25344&tenant=MT_SNY_9011